CLINICAL TRIAL: NCT05029037
Title: High-dose Intravenous Vitamin C (HDIVC) as Adjuvant Therapy in Critical Patients With Positive COVID-19. A Pilot Randomized Controlled Dose-comparison Trial.
Acronym: HDIVC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hugo Galindo (Other)
Responsible Party: Sponsor-Investigator, Hugo Galindo, Dr. Hugo Galindo, Fundacion Epheta
Organization: Fundacion Epheta (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAVCI
Record Dates: First submitted 2021-08-27; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: Vitamin C- Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 80 patients randomized to group A will receive two doses (High) of vitamin C intravenously, twice a day for seven days.
  Interventions: Drug: High doses of intravenous vitamin C
- Group B (Placebo Comparator): 80 patients assigned to group B will receive two doses of Dextrose 500 mL, twice a day for seven days.
  Interventions: Drug: Dextrose 500 mL

INTERVENTIONS:
Drug: High doses of intravenous vitamin C — Two (2) High doses of intravenous vitamin C for seven (7) days.
  Arms: Group A
Drug: Dextrose 500 mL — Application of a vial of LEV in 100 mL of water for injection, which is diluted in 400mL of 5% Dextrose for a final volume of 500mL of intravenous fluids, to be applied to the chosen patient, in a drip of 0.5 grams of the placebo solution per minute, for a total of 60 minutes.
  Twice a day for seven days.
  Arms: Group B

SUMMARY:
The objective of this study is to evaluate the impact of this HDIVC therapy in the first treatment of symptomatic Covid-19 patients in a time period of one week.

DETAILED DESCRIPTION:
We consider that treatment with high doses of injectable vitamin C HDIVC could have a positive impact as an adjunct on the immunity of patients with Covid while reducing the possibility of worsening their clinical picture. Similarly, we wish to evaluate the efficacy of this treatment, for one week, in patients hospitalized in the ICU, in order to reduce the inflammatory burden and reduce hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with consent, adult men or women, age ≥ 18 years.
* Laboratory confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assays; and/or clinical findings suggesting infection.
* Hospitalized with a SARS-CoV-2 infection of any duration.
* Ability to provide an informed consent signed by the study patient or a legally acceptable representative.
* Willingness and ability to comply with the procedures/evaluations related to the study.
* Have an oxygen saturation (SaO2) of 94% or less while breathing room air; or a ratio between the partial pressure of oxygen (PaO2) and the fraction of inspired oxygen (FiO2) (Pao2: Fio2) equal to or less than 300 mg. Hg. (WHO defines PAFI less than or equal to 250; being mild: 200-300; moderate: 100-200; severe: 100 or less.
* Normal kidney function: (creatinine 0.7 mg / dl for men or 20 to 200ng / ml and 0.6 to 1.1 mg / dl for women or 15-150 ng / ml); urinary output greater than or equal to 1 cc / kg / hour; glomerular filtration rate greater than 30 cc / min).
* Without chronic kidney disease (CKD) defined by stage II or higher according to the Kidney Disease Improving Global Outcomes (KDIGO) classification.

Exclusion Criteria:

* Age <18 or pregnant or lactating woman.
* Allergy to vitamin C.
* Severe liver failure.
* eGFR ≤ 30 ml / min / 1.73 m2 (defined by the CKD-EPI SCr formula).
* History of any organ transplants requiring treatment active immunosuppressant that may interfere with kidney function.
* If you required cardiopulmonary resuscitation (CPR) within 14 days, and/or DNR orders (do not resuscitate) DNI (do not intubate).
* If death is considered imminent or unavoidable during this admission, and the treating physician, patient, or surrogate decision-maker is not engaged in active treatment.
* Be on dialysis (either acute or chronic) or need dialysis imminent at the time of enrollment.
* Patients with known HIV infection.
* Patients with a known or suspected history of nephropathy due to oxalate or hyperoxaluria, scurvy, chronic iron overload, deficiency by G-6PD.
* Patients with known hemochromatosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Mean change in worst (highest) | Seven (7) days after randomization.
  Mean change in worst (highest) oxygenation level (oxygen saturation or oxygen flow in liters/min) in non-ventilated patients.
Mean change in worst (lowest) | Seven (7) days after randomization.
  Mean change in worst (lowest) PaO2 / FiO2 ratio (in mmHg) in ventilated patients. It should be within the first seven days after randomization.

SECONDARY OUTCOMES:
Mortality | up to day 28
  Mortality
Duration of mechanical ventilation | Days
  Duration of mechanical ventilation

IPD SHARING:
Plan to Share IPD: No